CLINICAL TRIAL: NCT04538924
Title: Multimodality Study on Etiologic Mechanisms, Myocardial Changes, and Prognosis of Patients With Myocardial Infarction With Non-obstructive Coronary Arteries
Brief Title: Etiologic Mechanisms, Myocardial Changes and Prognosis of Patients With MINOCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Research Council of Lithuania (Other)
Responsible Party: Principal Investigator, Rokas Šerpytis, Principal Investigator; MD, Vilnius University Hospital Santaros Klinikos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2MI-1
Record Dates: First submitted 2020-08-27; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Infarction With Nonobstructive Coronary Arteries
MeSH Terms: conditions — MINOCA | interventions — Laboratories

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINOCA (group I) - conventional MI treatment (Other): Traditional MI treatment with optimal doses of statin, angiotensin-converting enzyme inhibitors (ACEI) or angiotensin II receptor blockers (ARB), beta-blockers (BB) and dual antiplatelet therapy (DAPT).
  Interventions: Other: extended clinical, laboratory and instrumental examination; treatment options comparison
- MINOCA (group II) (Other): Treatment with a low-dose statin and ACEI/ARB. In case of vasospasm, calcium channel blockers.
  Interventions: Other: extended clinical, laboratory and instrumental examination; treatment options comparison

INTERVENTIONS:
Other: extended clinical, laboratory and instrumental examination; treatment options comparison — Multimodality investigation and different treatment comparison

SUMMARY:
This prospective trial will include 150 patients with myocardial infarction with non-obstructive coronary arteries (MINOCA). A thorough clinical, laboratory and imaging evaluation will be performed by novel biomarkers and modern imaging techniques (heart magnetic resonance imaging and noninvasive testing). Moreover, two different treatment groups will be distinguished. Additionally, a retrospective analysis of patients meeting MINOCA criteria will be performed.

DETAILED DESCRIPTION:
Primary goals The primary trial goal is to assess the etiologic mechanisms of myocardial damage in patients with MINOCA as well as to evaluate a variety of therapeutic strategies for these patients.

Secondary goals

1. To assess functional and morphological myocardial changes in patients with MINOCA;
2. To assess the true prevalence and prognostic relevance of MINOCA (all-cause mortality and MACE);
3. To test the effect of conventional acute MI therapies (BB, ACEI, ARB, CCB, statins, anti-platelet agents) on MACE (death and myocardial infarction) and all-cause mortality in patients with MINOCA;
4. To test the diagnostic and prognostic role of several biomarkers (sST2, BNP, cTnI, CRP, copeptin, procalcitonin, MR-proADM, galectin-3) in patients with MINOCA;
5. To assess the impact of MINOCA with respect to chronic health status, such as persistent angina symptoms, impairment in quality of life, and depression;
6. To evaluate systemic microcirculation status and assess its effect on long term outcomes.
7. To evaluate hospital mortality and all-cause death within 6 and 12 months follow-up;
8. To determine recurrent hospitalizations within 30-days, 6 and 12 months follow-up;
9. To assess peak creatine kinase, creatine kinase-MB and troponin levels during hospital stay;
10. To determine quality of life at 6 and 12 months assessed using the Euroqol 5D (EQ-5D) questionnaire (www.euroqol.org).

ELIGIBILITY:
Inclusion Criteria:

1. acute MI:

   * detection of a rise and/or fall of cardiac troponin(cTn) values with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following:
   * symptoms of acute myocardial ischaemia;
   * new ischaemic ECG changes;
   * development of pathological Q waves;
   * imaging evidence of new loss of viable myocardium or new regional wall motion abnormality in a pattern consistent with an ischaemic aetiology
2. non-obstructive coronary arteries on angiography:

   - the absence of obstructive coronary artery disease (CAD) on angiography, (i.e. no coronary artery stenosis ≥50%), in any potential infarct-related artery;

   This includes both patients with:
   * normal or near normal coronary arteries (no stenosis >30%)
   * mild coronary atheromatosis (stenosis >30% but <50%).
3. angiography performed within 24 - 48 hours
4. age >18 years
5. informed consent

Exclusion Criteria:

* acute kidney failure
* stage 4-5 chronic kidney disease
* contraindications for coronary angiography or CMR
* patients involved in another biomedical trial
* inability to make a decision to participate in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality | 12 months follow-up
Rate of cardiovascular death | 12 months follow-up

SECONDARY OUTCOMES:
Rate of hospitalization for MI | 12 months follow-up
Rate of MACE | 12 months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serpytis R, Majauskiene E, Navickas P, Lizaitis M, Glaveckaite S, Rucinskas K, Petrulioniene Z, Valeviciene N, Samalavicius RS, Berukstis A, Baranauskas A, Gargalskaite U, Laucevicius A, Chen QM, Alpert JS, Serpytis P. Randomized Pilot Trial on Optimal Treatment Strategy, Myocardial Changes, and Prognosis of Patients with Myocardial Infarction with Nonobstructive Coronary Arteries (MINOCA). Am J Med. 2022 Jan;135(1):103-109. doi: 10.1016/j.amjmed.2021.08.023. Epub 2021 Sep 22. PMID 34562410